CLINICAL TRIAL: NCT05004974
Title: Sintilimab Combined With Pemigatinib in Patients With PD-L1-positive and FGFR Mutated Advanced Non-small Cell Lung Cancer: an Open Label, Phase II Trial
Brief Title: Sintilimab With Pemigatinib in Patients With PD-L1-positive and FGFR Mutated Advanced Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K2021085
Record Dates: First submitted 2021-07-13; First posted 2021-08-13 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Advanced Non Small Cell Lung Cancer
MeSH Terms: interventions — sintilimab; pemigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab with Pemigatinib (Experimental): Sintilimab combined with Pemigatinib every 3 weeks (Q3W): Sintilimab is administered every 3 weeks (200mg, IV), Pemigatinib 13.5 mg once daily (QD) orally, continuous administration.
  Interventions: Drug: Sintilimab; Drug: Pemigatinib

INTERVENTIONS:
Drug: Sintilimab — Sintilimab is administered every 3 weeks (200mg, IV).
Drug: Pemigatinib — Pemigatinib 13.5 mg once daily (QD) orally, continuous administration.

SUMMARY:
Lung cancer is the leading cause of death from cancer in China. In recent years, immune checkpoint inhibitor has gradually become a research hotspot, and it has continuously achieved huge breakthroughs. The FDA and NMPA have approved multiple PD-1/PD-L1 inhibitors for first-line or second-line treatment of advanced or metastatic NSCLC. But In clinical practice, there is still some controversy about PD-1 inhibitor monotherapy, especially for patients with low PD-L1 expression, the efficacy of monotherapy needs to be further improved. Strong genetic and functional evidence indicates that FGFR dysregulation can lead to the development and progression of cancer. Genetic alterations of FGFR1, FGFR2 and FGFR3 have been found in a variety of tumors. Squamous non-small cell lung cancer has about 13% of FGFR variants, while there are only 4% of any FGFR variants in lung adenocarcinoma. Studies of FGFR inhibitors in NSCLC show that AZD4575 has shown partial efficacy in FGFR partially mutated and expanded lung squamous cell carcinoma. FGFR pathway is involved in the regulation of the tumor immune microenvironment. In the tumor suppressor model of rectal cancer, it has been observed that FGFR2 overexpression promotes the expression of PD-L1 by activating JAK/STAT3 pathway, leading to tumor growth. In a lung cancer suppressor mouse model, the combination of FGFR inhibitor and PD-1 inhibitor can improve tumor remission and prolong survival. Based on the preliminary clinical data, this study assumes that Sintilimab(anti-PD-1) combined with Pemigatinib(FGFR inhibitor) can further improve efficay of advanced NSCLC with PD-L1 positive and FGFR1-3 mutation) including but not limited to FGFR amplification, rearrangement/fusion, mutation, etc.).

DETAILED DESCRIPTION:
This study is a prospective, Phase II clinical study. 20 Histologically confirmed NSCLCs with unresectable or locally advanced, recurrent or metastatic disease not suitable for radical concurrent chemo-radiotherapy, treatment naive, and confirmed PD-L1 positive with FGFR 1-3 mutations are enrolled. The participants will receive Sintilimab combined with Pemigatinib every 3 weeks (Q3W): Sintilimab is administered every 3 weeks (200mg, IV), Pemigatinib 13.5 mg once daily (QD) orally, continuous administration. The subject will continue treatment until disease progression, intolerable toxicity, withdrawal of informed consent, start of other anti-tumor treatments, death or other conditions that should be stopped as prescribed by the protocol. The longest administration time of Sintilimab is 2 years (35 cycles). In consideration of the safety of the combination therapy, this study will conduct safety monitoring on the 6 subjects initially enrolled in the safety observation period (defined as 21 days after the subjects received the study drug treatment for the first time) . After the study enrollment reaches 6 subjects, enrollment will be suspended until the safety observation period of the 6th patient is over and the conditions for continuing the study are met. If ≥2 dose-limiting toxicity (DLT) are observed in these 6 patients, the investigators will review the data and discuss, and decide to revise the dosing regimen of the follow-up study to reduce the incidence of adverse events, or terminate it completely. If DLT is less than or equal to 1 of the 6 participants, the study will continue to follow the original protocol. The primary endpoint is objective response rate, the secondary endpoints are progression free survival, duration of response, time to response, disease control rate, overall survival, safety and tolerance.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Patients confirmed by histology or cytology non-small cell lung cancer with stage IIIB-IIIC and stage IV (UICC and AJCC, 8th edition TNM staging) which is unresectable or unsuitable for radical concurrent radiochemotherapy;
3. Not applicable to EGFR/ALK/ROS1 targeted therapy;
4. Histologically confirmed PD-L1 positive (TPS≥1%);
5. Histology confirmed FGFR1-3 mutations, including but not limited to amplification, mutation, fusion/rearrangement, etc.;
6. According to RECIST v1.1 version, there is at least one measurable lesion.
7. Not received any systemic anti-tumor therapy for advanced/metastatic diseases. For participants who have received adjuvant/neoadjuvant therapy, or have received radical radiochemotherapy for locally advanced disease, if the interval between disease progression or recurrence and the end of the last treatment is more than 6 months, these participants are allowed to be included in this study;
8. Not used small molecule multi-target inhibitors (including Anlotinib, Lenvatinib, Sorafenib, etc.) that target the FGFR pathway;
9. Have not previously received the following immune checkpoint inhibitor therapy: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or targeting another stimulating or synergistic inhibition of T cell receptors (including but not limited to CTLA-4 , OX-40, CD137, etc.);
10. ECOG physical status is 0-1;
11. Expected survival time> 3 months;
12. The participants are allowed to receive palliative radiotherapy (including craniocerebral radiotherapy for symptomatic brain metastases), but the radiotherapy must be completed at least 2 weeks before the first study drug is administered (the end of palliative radiotherapy for the central nervous system should be 4 weeks before the first study drug administration), and the radiotherapy-related toxicity is restored to less than or equal to 1 degree (CTCAE 5.0, except for hair loss), no corticosteroid treatment is required, and radiation pneumonia is confirmed to be excluded;
13. Sufficient organ function, participants need to meet the following laboratory indicators:

    1. The absolute value of neutrophils (ANC) ≥1.5x10^9/L when no granulocyte colony stimulating factor is used in the past 14 days;
    2. Platelets ≥100×10^9/L in the case of no blood transfusion in the past 14 days, ;
    3. Hemoglobin>9g/dL without blood transfusion or erythropoietin in the past 14 days ;
    4. Total bilirubin≤1.5 upper limit of normal (ULN); or total bilirubin>1.5 ULN but direct bilirubin≤1.0 ULN;
    5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) are ≤2.5 ULN (patients with liver metastases are allowed to have ALT or AST ≤5 ULN);
    6. Serum creatinine ≤1.5 ULN and creatinine clearance rate (calculated by Cockcroft-Gault formula) ≥50 ml/min;
    7. Good coagulation function, defined as the international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 ULN; if the participant is undergoing anticoagulation therapy, as long as the PT is within the proposed range of anticoagulant drugs;
    8. Normal thyroid function is defined as thyroid stimulating hormone (TSH) within the normal range. If the baseline TSH is outside the normal range, participants whose total T3 (or FT3) and FT4 are within the normal range can also be included;
    9. Myocardial enzyme spectrum is within the normal range (for example, simple laboratory abnormalities that are judged by the investigator to be of no clinical significance are also allowed to be included in the group);
14. For female participants of childbearing age, a urine or serum pregnancy test should be performed within 3 days before receiving the first study drug administration (day 1 of cycle 1)and the result should be negative . If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required. Women of non-bearing age are defined as at least 1 year after menopause, or have undergone surgical sterilization or hysterectomy;
15. If there is a risk of conception, all participants (whether male or female) need to use contraceptive measures with an annual failure rate of less than 1% during the entire treatment period until 120 days after the last study drug administration.

Exclusion Criteria:

* Exclusion criteria related to diseases or comorbidities:

  1. Diagnosis of other malignant diseases other than non-small cell lung cancer within 5 years before the first administration (excluding radically cured skin basal cell carcinoma, skin squamous epithelial carcinoma and/or radically excised carcinoma in situ);
  2. Currently participating in interventional clinical research treatment, or received other research drugs or used research devices within 4 weeks before the first administration;
  3. Received anti-tumor drug treatment (including Chinese herbal medicine with anti-tumor indications) within 28 days before using the first administration;
  4. Before starting treatment, have not fully recovered from toxicity and/or complications caused by any intervention (ie, ≤ Grade 1 or reached baseline, excluding fatigue or hair loss) ;
  5. Meningeal metastasis/cancerous meningitis or central nervous system metastasis with known symptoms. For asymptomatic participants or participants with stable brain metastases after local treatment, those participants are also allowed to join the group if the following conditions are met :1) There are measurable lesions outside the central nervous system; 2) No symptoms of the central nervous system or no aggravation of symptoms within at least 2 weeks; 3) There is no evidence of imaging progress at least 4 weeks before the first administration; 4) Those who do not need glucocorticoid therapy or stop glucocorticoid therapy within 14 days before the first study drug administration;
  6. There is clinically uncontrollable pleural effusion/abdominal effusion (patients who do not need to drain the effusion or stop drainage for 3 days without a significant increase in effusion can be included);
  7. Known human immunodeficiency virus (HIV) infection history or confirmed positive immunological test results;
  8. Acute or chronic active hepatitis B (defined as HBsAg positive and the HBV-DNA copy number is greater than the upper limit of the normal value of the laboratory department of the research center), active hepatitis C (HCV) infection (defined as HCV antibody positive and Patients whose HCV-RNA level is higher than the lower limit of detection), or patients with both hepatitis B surface antigen (HbsAg) and anti-HCV antibody positive at the same time. Note: Hepatitis B participant who meet the following criteria can also be included in the group:1) Before the first administration, the HBV viral load is less than 1000 copies/ml (200 IU/ml), and the participant should receive anti-HBV treatment during the entire study drug treatment period to avoid viral reactivation 2) For participants with anti-HBc (+), HBsAg (-), anti-HBs (-) and HBV viral load (-), there is no need to receive preventive anti-HBV treatment, but close monitoring of virus reactivation is required.
  9. There are any serious or uncontrollable systemic diseases, including:1) Clinically significant or uncontrolled heart diseases, including: uncontrolled arrhythmia (pacemaker is allowed or those with atrial fibrillation and well-controlled heart rate); resting electrocardiogram indicated major abnormalities with severe symptoms that are difficult to control in rhythm, conduction or morphology , such as complete left bundle branch block, heart block above Ⅱ degree, ventricular arrhythmia or atrial fibrillation; unstable angina, acute myocardial infarction, congestive heart failure, chronic heart failure of New York Heart Association (NYHA) grade ≥ 2 within 6 months before the first administration; 2) There are ECG changes or medical history that the investigator considers to be clinically significant; QTcF interval> 480 ms, for participants with indoor conduction block (QRS interval> 120 ms), JTc interval can be used instead of QTc interval (If JTc is used instead of QTc, JTc must be ≤340 ms); 3) Uncontrollable hypertension, systolic blood pressure> 160 mmHg or diastolic blood pressure> 100 mmHg after the best medical treatment, history of hypertensive crisis or hypertensive encephalopathy; 4) There is a serious infection in the active phase or poor clinical control; 5) There is clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction; 6) Liver diseases such as decompensated liver disease, hepatic encephalopathy, hepatorenal syndrome or Child-Pugh Class B and more severe liver cirrhosis, acute or chronic active hepatitis; 7) Poor control of diabetes (fasting blood glucose (FBG)> 10mmol/L); 8) Urine routines suggest that urine protein is ≥++, and the 24-hour urine protein quantitation is confirmed to be greater than 1.0 g;
  10. Have received a major surgical operation (except for surgery for the purpose of biopsy) within 4 weeks before the first administration or are expected to undergo major surgery during the study treatment;
  11. Before starting treatment, have not fully recovered from toxicity and/or complications caused by any intervention (such as major surgery) (ie, ≤ Grade 1 or reached baseline, excluding fatigue or hair loss); Exclusion criteria related to sintilimab treatment
  12. Have received systemic systemic treatment with anti-lung cancer Chinese patent medicines or immunomodulatory drugs (including thymosin, interferon, interleukin, except for local use to control pleural fluid) within 2 weeks before the first administration;
  13. An active autoimmune disease that requires systemic treatment (such as the use of disease-relieving drugs, glucocorticoids, or immunosuppressive agents) occurred within 2 years before the first administration. Alternative therapies (such as thyroxine, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency, etc.) are not considered systemic treatments;
  14. Are receiving systemic glucocorticoid therapy (excluding nasal spray, inhaled or other local glucocorticoids) or any other form of immunosuppressive therapy within 7 days before the first administration of the study; Note: The use of physiological doses of glucocorticoids (≤10 mg/day prednisone or equivalent drugs) is allowed;
  15. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
  16. A history of non-infectious pneumonia requiring glucocorticoid therapy within 1 year before the first administration, or current clinically active interstitial lung disease;
  17. Active tuberculosis;
  18. Live vaccine has been vaccinated within 30 days before the first administration (cycle 1, day 1); Note: It is allowed to receive inactivated virus vaccine for seasonal influenza within 30 days before the first administration; however, it is not allowed to receive live attenuated influenza vaccine for intranasal administration.

      Exclusion criteria related to Pemigatinib:
  19. Have received selective FGFR inhibitor treatment in the past;
  20. A history of disorder of calcium and phosphorus metabolism or systemic electrolyte metabolism imbalance with ectopic soft tissue calcification (except for skin, kidney, tendon, or blood vessel calcification caused by injury, disease, and advanced age without systemic electrolyte metabolism imbalance) ；
  21. The following laboratory parameters are abnormal:1) Serum phosphate>1.0 ULN; 2) Serum calcium is out of the normal range, or when the serum albumin is out of the normal range, the corrected calcium concentration of serum albumin is out of the normal range; 3) Potassium level <lower limit of normal value; Potassium level can be corrected by supplements during screening.
  22. Corneal or retinal disease confirmed by ophthalmological examination as having clinical significance;
  23. Any strong CYP3A4 inhibitors or inducers have been used within 14 days or 5 half-lives (whichever is shorter) before the first administration of the study drug. Allow topical ketoconazole;
  24. People with multiple factors that affect oral medications (such as inability to swallow, gastrointestinal resection, significant digestive system diseases that may interfere with absorption, metabolism, or excretion, such as chronic diarrhea or intestinal obstruction, etc.);
  25. The participant has a history of vitamin D deficiency and requires super-physiological supplementation of vitamin D (except for vitamin D dietary supplements).

      Other:
  26. Those who are known to be allergic to Sintilimab, Pemigatinib and their active ingredients or excipients;
  27. Pregnant or lactating women, or participants who are expected to conceive or give birth during the study period from the screening visit to the completion of the safety follow-up visit (male participants to 90 days after the last dose);
  28. Other acute or chronic diseases, mental illnesses, or abnormal laboratory test values that may cause the following results: increase the risk related to study participation or study drug administration, or interfere with the interpretation of study results, and the patients not eligible to participate in this study judge by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 6 weeks
  The proportion of subjects who achieved complete remission (CR) or partial remission (PR) according to the RECIST1.1.

SECONDARY OUTCOMES:
Progression-free survival | 9 months
  the time from first administration to disease progression or death
Duration of remission | 6 months
  the time from the date of the first CR or PR to PD, and is only used for subjects who have achieved objective remission
Time to remission | 6 weeks
  the time from the first administration to the first CR or PR, and is only used for patients who have achieved objective remission
Disease control rate | 6 weeks
  Proportion of subjects with CR, PR and stable disease
Overall survival | 4 years
  Time from first administration to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Affiliated Hospital of Zhejiang University, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No